CLINICAL TRIAL: NCT04863118
Title: Acute Effects of Strength Training in Shallow Water and Dry Land and High-intensity Training in Shallow and Deep Water, on Functional Measures and Biochemistries of Individuals With Parkinson's Disease
Brief Title: Acute Effects of Strength Training and High Intensity Training on Functional and Biochemical Measurements of Individuals With Parkinson's Disease in Different Environments and Depths
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Fernanda Cechetti, Clinical Professor, Ph.D, Fernanda Cechetti, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: DPEAQ21
Record Dates: First submitted 2021-04-11; First posted 2021-04-28 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Parkinson Disease and Hydrotherapy
Keywords: Parkinson's disease; Physiotherapy; Hydrotherapy; Gait; Posture
MeSH Terms: conditions — Parkinson Disease | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strength training protocol performed in shallow water and dry land (Experimental): Parkinson Disease and healthy individuals
  Interventions: Other: Strength training in shallow water and dry land
- High-intensity training protocol performed in shallow and deep water (Experimental): Parkinson Disease and healthy individuals
  Interventions: Other: High-intensity training in shallow and deep water

INTERVENTIONS:
Other: Strength training in shallow water and dry land — Dry land: The intervention will last for 60 minutes, consisting of exercises to strengthen the global extensor musculature, that is, involving the upper limbs, trunk and lower limbs. Weights and equipment for strength training will be used. The sessions will start with 10 minutes of warm-up, the central part of exercises to strengthen the extensor muscles and the last part will consist of oriented stretches. In the central part, a typical strength training will be performed (2-6 series; 85% of RM), using submaximal subjective effort and with repetition control.
  Shallow water: The intervention performed on dry land will be adapted and produced in an aquatic environment. Aquatic implements will be used for strength training.
  Arms: Strength training protocol performed in shallow water and dry land
Other: High-intensity training in shallow and deep water — Shallow water: The intervention will last 60 minutes. The exercises consist of: immersion, balance, strength, agility and displacement in the water. As they will start with 10 minutes of warm-up and the last part will consist of stretches oriented along the edge of the pool and on the depth reduction platform. In the main part of the intervention, different styles of exercises will be performed, with or without the use of implements. Displacements will have varying speeds in the same session, defined by Borg's Scale of subjective sensation of effort.
  Deep water: The intervention carried out in shallow water will be adapted with the use of floating belts and reproduced in deep water.
  Arms: High-intensity training protocol performed in shallow and deep water

SUMMARY:
Introduction: Parkinson's disease (PD) is the second most common neurodegenerative disease in the elderly. Chronic and progressive, it includes loss of dopamine, a neurotransmitter involved in the regulation of movement. Thus, functional changes, such as postural disorders, trunk flexor pattern, muscle activation deficits, impairment of gait, balance, and mobility are common findings in this population. Once there is dopaminergic depletion, it is important to identify mechanisms that act in the production and survival of nigral dopaminergic neurons, like the brain-derived neurotrophic factor (BDNF). Studies describe a correlation between serum BDNF levels and PD motor dysfunction. Still, it is presumed that physical therapy can positively regulate substances that act directly on the Central Nervous System, such as BDNF. Physical exercise, in addition to promoting biochemical modulations in PD, can provide benefits in motor symptoms that sometimes do not improve with drugs. Conventional physiotherapy performed on dry land is a therapeutic resource used in PD. The conventional physiotherapy is useful for management of functional changes caused by PD due to muscle strengthening exercises. These exercises can be adapted and performed in water, at different depths, shallow and deep water. Thus, aquatic physiotherapy has been shown to be able to interfere in PD motor disorders, with perspective of maximizing the rehabilitation program effects due to the physical properties of water. These reasons, in addition to the large use of these interventions in the clinical practice and their likely benefits in the PD alterations, suggest the importance of studies in this area. Furthermore, the immediate effects of strengthening interventions with global extensor musculature emphasis on global extensor musculature, and of high-intensity training protocols, which encompass different environments and different depths, on functional and biochemical measures of PD are poorly studied.

Objectives: To verify the acute effects of a global extensor musculature strength training protocol, performed on dry land and shallow water, and of a high-intensity training protocol performed in shallow and deep water on functional and biochemical measurements of individuals with PD.

Methods: This will be a single-blind crossover, cross-sectional study with a 24-hour follow-up. The sample will be composed of subjects between 50 and 70 years old, classified from 1 to 3 in the Hoehn and Yahr scale, with a PD diagnosis rigid-akinetic and/or tremor-dominant type in the "OFF" period of the medication. In this research there will be an intervention group (IG) composed of individuals with Parkinson's disease and a control group (CG) of healthy individuals. Both will be randomly distributed in a randomized way and submitted to two different training sessions, for 60 minutes, at different times, in order to analyze the acute effects and follow-up of the following interventions: a strength training of the global extensor musculature in dry land and shallow water (120 cm deep) and high-intensity training (Borg Scale), at different depths: shallow water (120 cm deep) and deep water. To characterize the sample, anamnesis and Motor Examination of Movement Disorder Society Unified Parkinson Disease Rating Scale (MDS-UPDRS III) will be performed. The individuals will be submitted to pre, post and 24h evaluations after the intervention. Functional measures will be analyzed: postural stability, by stabilometry; strength, by isokinetic dynamometry; spatiotemporal gait variables, with kinematic analysis; balance, with Berg Balance Scale and functional mobility with Timed Up and Go test and biochemical analysis: venous blood collection and ELISA test will be performed measuring serum BDNF levels. In this way, the acute effects of the global extensor musculature strength training protocol and of high-intensity training on the different variables analyzed, environments, depths and moments of evaluation will be analyzed and compared.

ELIGIBILITY:
Inclusion Criteria:

GI (Individuals with Parkinson Disease):

* Individuals diagnosed with Parkinson's disease for at least 6 months;
* Age between 50 to 70 years;
* Classified on the Hoehn and Yahr scale from 1 to 3;
* Rigid-akinetic and/or tremor-dominant type;
* Individuals who have preserved their cognitive skills, assessed by means of the Mini Mental State Examination (MMSE) and who have a cut-off score of 23/24 (FOLSTEIN et al., 1975).

GC (Healthy individuals):

* Age between 50 to 70 years;
* Individuals who have preserved their cognitive skills (with the same cut-off score as the GI in the MMSE);
* Walk independently.

Exclusion Criteria:

GI (Individuals with Parkinson Disease):

* Individuals who have other associated musculoskeletal and neurological disorders;
* Individuals with dementia installed;
* Individuals with pathologies and injuries associated with the skin that make it impossible to enter the aquatic environment;
* Individuals with hydrophobia.

GC (Healthy individuals):

* Individuals who have musculoskeletal and neurological pathologies;
* Individuals with dementia installed;
* Individuals with pathologies and injuries associated with the skin that make it impossible to enter the aquatic environment;
* Individuals with hydrophobia.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Changes in postural stability (stabilometry) | Changes between pre and post immediate intervention. Changes 24 hours after interventions.
  Stabilometry will be used as a method of evaluating the postural balance of the analyzed subjects by quantifying their oscillations, thus, measurements of the levels of stability will be performed when standing in an upright position, with eyes open and closed. Data will be collected through the AMTI force platform - OR6-6 Force plate with MAS-6 amp. The patient will be positioned in an upright posture on the platform, as relaxed as possible, with barefoot and approximately shoulder width apart as described by Laufer; Ashkenazi and Josman (2008). The subject will be asked to look at a point fixed to a wall in front of him, at eye level. Three attempts will be made with an initial 20 seconds for adaptation that will be discarded followed by 25 seconds of valid collection.

SECONDARY OUTCOMES:
Strength (isokinetic dynamometry) | Changes between pre and post immediate intervention. Changes 24 hours after interventions.
  Isokinetic dynamometry aims to assess an individual's muscle condition, measuring their strength, power and endurance, determining the degree of muscle deficiency they present. The individuals will be submitted to an assessment of the isometric torque in flexion and maximum extension of upper limbs, trunk and lower limbs using the Cybex Norm isokinetic dynamometer (Cybex Inc., Ronkonkoma, NY, USA). For familiarization, there will be two submaximal isometric contractions in each position. The evaluation protocol consists of three maximum voluntary isometric contractions, lasting 5 seconds in each position. Participants will be verbally encouraged during contractions, with an interval of 2 minutes between each contraction, to avoid fatigue. An interval of 20 minutes will be made between the assessments of the flexion torque for the extension of the upper limbs, trunk and lower limbs. The contraction with the highest torque value will be applied for data analysis using the Humac software
Spatiotemporal gait variables (kinematic analysis) | Changes between pre and post immediate intervention. Changes 24 hours after interventions.
  For the kinematic analysis, 22 reflective markers will be positioned on both sides of the body in order to use a modified full body model that the program uses. A treadmill will be used for the tests. 3D kinematic data will be collected from image records using a VICON kinematics system, which consists of six synchronized cameras that use a shooting frequency of 100 Hz. After system calibration and placement of markers, the acquisition phase where each participant will be guided and positioned on a force platform and instructed to maintain an orthostatic position with the feet aligned, during a period of 5 seconds for system calibration. Next, gait assessment will be carried out, where the subjects will have to walk independently, as usual, with barefoot, on a specific path on a 8m long and 1.4m wide walkway at a self-selected speed.
Balance (Berg's Balance Scale - BBS) | Changes between pre and post immediate intervention. Changes 24 hours after interventions.
  The BBS will be used to assess the static, dynamic balance and the risk of falls of the analyzed subjects. This scale assesses the performance of functional balance with 14 tests, which are directed to the individual's ability to sit, stand, reach, rotate around himself, look over his shoulders, stand in one-leg support and take steps. It has a maximum score of 56 points and a minimum of 0 points, where 17 each test has five alternatives ranging from 0 to 4 points (MIYAMOTO et al., 2004).
Functional mobility (Timed Up and Go test - TUG) | Changes between pre and post immediate intervention. Changes 24 hours after interventions.
  To assess functional mobility, the TUG will be performed, in which the subject starts sitting in a chair, walks for a distance of 3 meters, goes around a cone, returns and sits down on the chair again. The subject is oriented to perform the test as soon as possible. Free individuals and have less than 10 seconds, since they have reasonable balance and gait speed, while dependents have 30 seconds or more.
Biochemical analysis of the serum BDNF level (venous blood collection) | Changes between pre and post immediate intervention. Changes 24 hours after interventions.
  The biochemical measurements of the serum BDNF level will be analyzed by means of blood collection and ELISA test, blood samples (approximately 5 mL) will be collected between 7:00 am and 9:00 am, in the pre, post and 24h evaluation after the last session. The tubes will be centrifuged at 1048g for 10 min. Serum BDNF levels will be determined by the immunoenzymatic assay method (ELISA), with a specific kit (Promega, USA). All samples will be measured in duplicate by a SpectraMax M2e microplate reader (Molecular Devices, USA).
Biochemical analysis of the serum cortisol level (venous blood collection) | Changes between pre and post immediate intervention. Changes 24 hours after interventions.
  The biochemical measurements of the serum BDNF level will be analyzed by means of blood collection and ELISA test, blood samples (approximately 5 mL) will be collected between 7:00 am and 9:00 am, in the pre, post and 24h evaluation after the last session. The tubes will be centrifuged at 1048g for 10 min. Serum cortisol levels will be measured by Enzyme Immunoassay (EIA) according to the manufacturer's instructions (Accubind, USA). All samples will be measured in duplicate by a SpectraMax M2e microplate reader (Molecular Devices, USA).

CONTACTS AND LOCATIONS:
Locations (1):
- Fernanda Cechetti, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886